CLINICAL TRIAL: NCT02918799
Title: Pilot of Culturally Tailored Mpowerment for HIV Prevention Among YMSM in Beirut
Brief Title: Pilot of Mpowerment for Young Men Who Have Sex With Men (YMSM) in Beirut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Lebanese AIDS Society (Unknown); Arab Foundation for Freedom and Equality (Unknown); University of California, San Francisco (Other); AIDS Project Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-0992
Record Dates: First submitted 2016-09-16; First posted 2016-09-29 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Intervention will be evaluated with community cohort and use of pre- post-intervention analysis plan
Oversight: Data Monitoring Committee: No

ARMS (1):
- Community cohort (Other): Beirut community will receive the multi-component intervention Mpowerment; the community cohort of YMSM will be used to evaluate the effects of the intervention on the community, as the cohort participants may or may not have participated in the intervention.
  Interventions: Behavioral: Mpowerment

INTERVENTIONS:
Behavioral: Mpowerment — MP is a multi-level intervention that reaches out to all YMSM in a community by mobilizing men to encourage their friends to reduce risk behavior and join the program (informal outreach), along with holding social activities that promote safe sex (formal outreach). MP provides YMSM with skills, support and confidence to find solutions within themselves for sexual health, and seeks to affirm the validity and rights of same-sex behavior and identities.

SUMMARY:
This project will adapt and pilot a multi-level, community-based intervention to promote HIV prevention and sexual health among young men who have sex with men in Beirut.

DETAILED DESCRIPTION:
Mpowerment (MP) is an evidence-based community-level, structural, social and behavioral intervention for HIV prevention developed for YMSM that targets individual and community empowerment and mobilization, self-affirmation, sexual self-knowledge, and creation of a supportive social environment. MP has been widely used in the U.S., but not in a mostly Muslim setting. This project will adapt and pilot MP for the sociocultural issues facing YMSM (age 18-29) in Beirut. There will be a 2-year pilot implementation of MP, with longitudinal cohorts of YMSM in Beirut and Jounieh, the latter being the control community. Primary outcomes will be unprotected anal sex and HIV testing, with secondary outcomes being engagement in peer outreach, and perceived peer norms related to condom use and HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18-29, who have had anal sex with men in the past 6 months

Exclusion Criteria:

* not residing in Lebanon

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
condomless anal sex | past 3 months
  condomless anal sex with HIV+ or unknown status partners in past 3 months will be assessed via questionnaire
HIV testing | past 6 months
  Variable will be assessed via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, PhD, Principal Investigator — RAND

IPD SHARING:
Plan to Share IPD: No